CLINICAL TRIAL: NCT02883634
Title: Short, Medium and Long Term Effects of Specific and Nonspecific Spinal Manipulative Therapy in Patients With Chronic Non-specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Specific or Non-Specific Manipulation for Patients With Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Ronaldo Fernando de Oliveira, PhD Student, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNICID10
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Low Back Pain
Keywords: Back pain; spinal manipulation
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- specific manipulation (Experimental): Participants allocated to group "specific manipulation", will have their lumbar spine manipulated according to the previous clinical examination.
  Interventions: Other: Specific manipulation
- non-specific manipulation (Experimental): Participants allocated to group "non-specific manipulation" will have their upper thoracic spine manipulated (also known as "global manipulation") regardless of the previous clinical examination.
  Interventions: Other: Non-specific manipulation

INTERVENTIONS:
Other: Specific manipulation — Patients allocated to the specific manipulation group will receive spinal manipulation according to the physical examination performed prior to the treatment allocation.
  Arms: specific manipulation
Other: Non-specific manipulation — Patients allocated to the specific manipulation group will receive spinal manipulation on the upper thoracic spine that will be not related to the physical examination performed prior to the treatment allocation.
  Arms: non-specific manipulation

SUMMARY:
We aim to evaluate the long-term effects of 10 sessions of spinal manipulative therapy applied in a vertebral region-specific or region nonspecific level immediately after treatment and 3 and 6 months after randomization.

DETAILED DESCRIPTION:
To evaluate the long-term effects of 10 sessions of spinal manipulative therapy applied in a vertebral region-specific or region nonspecific level immediately after treatment and 3 and 6 months after randomization.

148 patients with chronic non-specific low back pain will be enrolled for this clinical trial. Patients will undergo to a specific physical examination in order to determine the ideal lumbar spine level to be manipulated. The outcomes of interest are pain intensity, pain pressure threshold, global perceived effect and disability associated with back pain. After the first assessment patients will be randomly assigned to two groups that will receive 10 sessions of spinal manipulation over a period of four weeks, and may receive manipulation according to the findings on physical examination (specific manipulation) or may receive manipulation in the upper thoracic region, disregarding the physical examination findings (nonspecific manipulation).

ELIGIBILITY:
Inclusion Criteria:

- Patients with low back pain duration from 3 to 24 months.

Exclusion criteria:

* Patients with a pain duration lower than 3 months and higher than 24 months.
* Patients with nerve root compromise or with serious spinal pathology,
* Pregnant patients,
* Previous back surgery
* Patients with any contra-indication to spinal manipulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks
  Pain intensity will be measured using a 0-10 numerical rating scale

SECONDARY OUTCOMES:
Pain Intensity | 3 and 6 months after randomization
  Pain intensity will be measured using a 0-10 numerical rating scale
Disability | 4 weeks, 3 and 6 months after randomization
  Disability will be measured by the 0-24 Roland Morris Disability Questionnaire
Global Impression of Recovery | 4 weeks, 3 and 6 months after randomization
  Global impression of recovery will be measured by an 11-item Global Perceived Effect Scale
Pressure Pain Threshold | 4 weeks after randomization
  Pressure Pain Threshold will be measure by a digital pressure algomoter

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Costa, PT, PhD, Study Chair — Universidade Cidade de São Paulo
Locations (1):
- Universidade Cidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We are happy to share our data with researchers that would like to use it on an IPD.

REFERENCES:
- [Derived] de Oliveira RF, Costa LOP, Nascimento LP, Rissato LL. Directed vertebral manipulation is not better than generic vertebral manipulation in patients with chronic low back pain: a randomised trial. J Physiother. 2020 Jul;66(3):174-179. doi: 10.1016/j.jphys.2020.06.007. Epub 2020 Jul 10. PMID 32660919